CLINICAL TRIAL: NCT03373344
Title: Remediation of Emotional Processing Deficits in MS: A Randomized Clinical Trial
Brief Title: Remediation of Emotional Processing Deficits in MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Responsible Party: Principal Investigator, Helen Genova, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R-920-16
Record Dates: First submitted 2017-12-08; First posted 2017-12-14 (Actual); Last update posted 2020-07-10 (Actual); Status verified 2020-07

CONDITIONS: Multiple Sclerosis
Keywords: emotional processing; multiple sclerosis; cognition
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants in the experimental group will receive emotional processing training exercises administered on a laptop computer. They will undergo 12 sessions of 45-60 minutes each (twice a week for 6 weeks).
  Interventions: Behavioral: Emotional Processing Training
- Control Group (Placebo Comparator): Participants in the control group will meet with the examiner the same frequency and for the same duration as those in the experimental group.
  They will receive placebo control exercises administered on a laptop computer.
  Interventions: Behavioral: Placebo control exercises

INTERVENTIONS:
Behavioral: Emotional Processing Training — Participants in the experimental group will receive computerized exercises administered on a laptop computer. They will undergo 12 sessions of 45-60 minutes each (twice a week for 6 weeks).
  Arms: Experimental Group
Behavioral: Placebo control exercises — Participants in the control group will receive computerized control exercises administered on a laptop computer. They will undergo 12 sessions of 45-60 minutes each (twice a week for 6 weeks).
  Arms: Control Group

SUMMARY:
This study will test the effectiveness of an emotional processing intervention in individuals with MS in a double blind placebo controlled randomized clinical trial. We will utilize an intervention which has been successfully used in other populations, including Schizophrenia and Traumatic Brain Injury. Our pilot data shows that this intervention is effective in individuals with MS as well

DETAILED DESCRIPTION:
This study will test the effectiveness of an emotional processing intervention in individuals with MS in a double blind placebo controlled randomized clinical trial RCT). We will utilize an intervention which has been successfully used in other populations, including Schizophrenia and Traumatic Brain Injury. Our pilot data shows that this intervention is effective in individuals with MS, as well.

All participants will undergo a baseline evaluation assessing emotional processing abilities, cognitive functioning, and psychological functioning. Participants will then be randomized into two groups. During the treatment phase, the experimental group will receive the proposed intervention while the control group will receive a "placebo" treatment. Neuropsychological assessment will be repeated at the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 18-65.
* diagnosis of Relapsing-Remitting Multiple Sclerosis.
* can read and speak English fluently.

Exclusion Criteria:

* history of prior stroke or other neurological disease or injury.
* history of significant psychiatric illness (for example, bipolar disorder, schizophrenia, or psychosis) or a current diagnosis of Major Depressive Disorder, Schizophrenia, Epilepsy, Bipolar Disorder.
* significant alcohol or drug abuse history.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Emotional Processing | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  Change in scores on computerized tests of emotional processing

SECONDARY OUTCOMES:
Emotional Function | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  Change in scores on self-report of emotional functioning, measured via questionnaire
Self report of Quality of Life | Scores will be assessed at two time-points, baseline (week 1) and post-intervention (week 8)
  Change in scores on self-report of quality of life, measured via questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Helen Genova, PhD, Principal Investigator — Research Scientist
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States